CLINICAL TRIAL: NCT01214226
Title: Evaluation of the Survival Benefit of the Adjunction of Pentoxifylline to Corticosteroids in Patients Suffering From Severe Alcoholic Hepatitis
Brief Title: Double-blind Randomized Controlled Trial in Severe Alcoholic Hepatitis
Acronym: CorpentoxHAA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Service des Maladies de l'Appareil Digestif, Hôpital Huriez,, CHRU Lille, France (Pr Philippe Mathurin / MD, PhD)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-006944-78; PROM 2006/0636 (Other: CHRU de Lille - promoteur); 2006-006944-78 (EudraCT Number)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-09

CONDITIONS: Alcoholic Hepatitis; Alcoholic Liver Disease
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxifylline + Prednisolone (Active Comparator): Pentoxifylline 400 mg prolonged-released tablets 3 time a day [1200 mg/day]
  + Prednisolone 2 ORODISPERSIBLE TABLETS OF 20 MG 1 TIME PER DAY [40 mg/day]
  Interventions: Drug: placebo
- Placebo + Prednisolone (Placebo Comparator): Placebo prolonged-release tabled 3 time a day
  + Prednisolone 2 ORODISPERSIBLE TABLETS OF 20 MG 1 TIME PER DAY [40 mg/day]
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — 400 mg prolonged-released tablets 3 time per day for 1 month.
  Other Names: TORENTAL 400MG
  Arms: Placebo + Prednisolone
Drug: placebo — prolonged-release tablets 3 time per day for 1 month
  Arms: Pentoxifylline + Prednisolone

SUMMARY:
The treatment of severe forms of alcoholic hepatitis (AH) constitutes a major challenge for clinicians involved in the management of severe alcoholic liver disease. In patients with Maddrey function higher than 32, compelling evidence from data has shown that corticosteroids improve short-term survival. However, novel strategies or molecules are required in light of the fact that approximately 40 % of patients continue to die at 6 months. A double-blinded randomized controlled trial of 101 patients has showed that Pentoxifylline improves survival of patients with severe AH, as compared to placebo. In terms of mechanisms, the effect of pentoxifylline is related to prevention of hepatorenal function whereas corticosteroids induce an early improvement in liver function. When considering these differences of mechanisms, many clinicians suggest that the addition of pentoxyfilline to corticosteroids is an attractive option that needs to be tested in patients with severe AH.

DETAILED DESCRIPTION:
The aim of the present study is to determine whether or not the adjunction of Pentoxifylline to corticosteroids would improve 6-month survival of patients with severe alcoholic hepatitis. This multicenter, randomized, double-blinded, controlled, phase 3 trial was conducted in 24 centers located in France and Belgium. Alcoholic hepatitis was biopsy-proven. All eligible patients were randomly assigned in a 1:1 ratio to receive corticosteroids + Pentoxifylline or corticosteroids + Placebo. The primary outcome of the study was 6-month survival. Assuming a two-sided type I error of 0.05, a randomization ratio of 1:1 between the 2 groups, 6-month survival of 64% in the Placebo and Corticosteroids group and of 78 % in the Pentoxifylline and Corticosteroids group, we estimated that with 268 randomized patients (134 in each group), the study would have a power of 80% to detect this increase in 6-month survival in the Pentoxifylline and Corticosteroid group.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol consumption more than 40 gram/day for women and 50 gram/day for men
* Maddrey discriminant function higher than 32
* Onset of jaundice within the 3 previous months
* Biopsy-proven alcoholic hepatitis

Exclusion Criteria:

* Hypersensitivity to pentoxifylline
* Any severe disease that may potential affect survival such as cardiac failure, ischemic cardiopathy, respiratory failure
* Any neoplasm that occurred within the 2 previous years
* Hepatocellular carcinoma or any previous diagnosis of hepatocellular carcinoma
* Portal thrombosis
* Severe gastrointestinal bleeding
* Uncontrolled sepsis within the 7 previous days
* Hepatorenal syndrome type I
* Viral and fungal infection
* Acute pancreatitis
* Any tuberculosis that occurred within the 5 previous years
* Psychiatric disorders that contraindicate the use of corticosteroids
* Infection related to virus of the hepatites B or C
* HIV infection (Human immunodeficiency virus)
* Any treatment with corticosteroids, immunosuppressive agents, budesonide, thalidomide or pentoxifylline that was given within the previous year
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 6 months

SECONDARY OUTCOMES:
Hepatorenal syndrome | 6 months
Score of Lille model | Seven days
Percentage of Meld score (Model for End-stage Liver Disease) higher than 17 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MATHURIN, MD PhD, Principal Investigator — University Hospital, Lille
Locations (28):
- University hospital, Brussels, Belgium
- France (27):
  - University hospital, Angers
  - Centre hospitalier, Béthune
  - Hôpital Jean Verdier (AH-HP), Bondy
  - University hospital, Bordeaux
  - University hospital, Caen
  - Hospital Antoine Béclère (Assistance Publique des Hôpiaux de Paris), Clamart
  - Hôpital Beaujon (AH-HP), Clichy
  - Centre Hospitalier, Creil
  - Hôpital Henri Mondor (AP-HP), Créteil
  - Centre hospitalier, Dunkirk
  - Centre Hospitalier, Lens
  - University hospital, Lille
  - Centre hospitalier Sambre en avesnois, Maubeuge
  - University hospital, Montpellier
  - University hospital, Nantes
  - University hospital, Nice
  - Hôpital Saint Antoine (AP-HP), Paris
  - Hôpital de la Pitié-Salpétrière (AP-HP), Paris
  - Hôpital Cochin (AH-HP), Paris
  - University hospital, Poitiers
  - University hospital, Rennes
  - Centre Hospitalier Victor Provo, Roubaix
  - University Hospital, Strasbourg
  - Centre Hospitalier, Tourcoing
  - Centre Hospitalier, Valenciennes
  - University hospital, Nancy, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse (AH-HP), Villejuif

REFERENCES:
- [Result] Lucey MR, Mathurin P, Morgan TR. Alcoholic hepatitis. N Engl J Med. 2009 Jun 25;360(26):2758-69. doi: 10.1056/NEJMra0805786. No abstract available. PMID 19553649
- [Result] Louvet A, Wartel F, Castel H, Dharancy S, Hollebecque A, Canva-Delcambre V, Deltenre P, Mathurin P. Infection in patients with severe alcoholic hepatitis treated with steroids: early response to therapy is the key factor. Gastroenterology. 2009 Aug;137(2):541-8. doi: 10.1053/j.gastro.2009.04.062. Epub 2009 May 13. PMID 19445945
- [Result] Louvet A, Naveau S, Abdelnour M, Ramond MJ, Diaz E, Fartoux L, Dharancy S, Texier F, Hollebecque A, Serfaty L, Boleslawski E, Deltenre P, Canva V, Pruvot FR, Mathurin P. The Lille model: a new tool for therapeutic strategy in patients with severe alcoholic hepatitis treated with steroids. Hepatology. 2007 Jun;45(6):1348-54. doi: 10.1002/hep.21607. PMID 17518367
- [Result] Mathurin P. Corticosteroids for alcoholic hepatitis--what's next? J Hepatol. 2005 Sep;43(3):526-33. doi: 10.1016/j.jhep.2005.06.003. No abstract available. PMID 16026887
- [Result] Naveau S, Chollet-Martin S, Dharancy S, Mathurin P, Jouet P, Piquet MA, Davion T, Oberti F, Broet P, Emilie D; Foie-Alcool group of the Association Francaise pour l'Etude du Foie. A double-blind randomized controlled trial of infliximab associated with prednisolone in acute alcoholic hepatitis. Hepatology. 2004 May;39(5):1390-7. doi: 10.1002/hep.20206. PMID 15122768
- [Result] Mathurin P, Abdelnour M, Ramond MJ, Carbonell N, Fartoux L, Serfaty L, Valla D, Poupon R, Chaput JC, Naveau S. Early change in bilirubin levels is an important prognostic factor in severe alcoholic hepatitis treated with prednisolone. Hepatology. 2003 Dec;38(6):1363-9. doi: 10.1016/j.hep.2003.09.038. PMID 14647046
- [Result] Mathurin P, Mendenhall CL, Carithers RL Jr, Ramond MJ, Maddrey WC, Garstide P, Rueff B, Naveau S, Chaput JC, Poynard T. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis (AH): individual data analysis of the last three randomized placebo controlled double blind trials of corticosteroids in severe AH. J Hepatol. 2002 Apr;36(4):480-7. doi: 10.1016/s0168-8278(01)00289-6. PMID 11943418
- [Result] Mathurin P, Duchatelle V, Ramond MJ, Degott C, Bedossa P, Erlinger S, Benhamou JP, Chaput JC, Rueff B, Poynard T. Survival and prognostic factors in patients with severe alcoholic hepatitis treated with prednisolone. Gastroenterology. 1996 Jun;110(6):1847-53. doi: 10.1053/gast.1996.v110.pm8964410.
- [Result] Ramond MJ, Poynard T, Rueff B, Mathurin P, Theodore C, Chaput JC, Benhamou JP. A randomized trial of prednisolone in patients with severe alcoholic hepatitis. N Engl J Med. 1992 Feb 20;326(8):507-12. doi: 10.1056/NEJM199202203260802. PMID 1531090
- [Derived] Mathurin P, Louvet A, Duhamel A, Nahon P, Carbonell N, Boursier J, Anty R, Diaz E, Thabut D, Moirand R, Lebrec D, Moreno C, Talbodec N, Paupard T, Naveau S, Silvain C, Pageaux GP, Sobesky R, Canva-Delcambre V, Dharancy S, Salleron J, Dao T. Prednisolone with vs without pentoxifylline and survival of patients with severe alcoholic hepatitis: a randomized clinical trial. JAMA. 2013 Sep 11;310(10):1033-41. doi: 10.1001/jama.2013.276300. PMID 24026598